CLINICAL TRIAL: NCT02363192
Title: The Effectiveness of Pharmacist Interventions in Improving Asthma Control and Quality of Life in Patients With Difficult Asthma
Brief Title: Effectiveness of Pharmacist Interventions in Difficult Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PH10/9328
Record Dates: First submitted 2015-02-09; First posted 2015-02-13 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Asthma
Keywords: Pharmacy
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pharmacist Intervention Group (Experimental)
  Interventions: Behavioral: Pharmacist intervention and pharmacist support
- Usual Care Group (No Intervention)

INTERVENTIONS:
Behavioral: Pharmacist intervention and pharmacist support — Patients randomised to this group will undergo an asthma assessment to assess asthma control, adherence and inhaler technique, by an Advanced Clinical Pharmacist specialising in Respiratory Medicine.
  Arms: Pharmacist Intervention Group

SUMMARY:
Of the 5.2 million people with asthma in the UK, approximately one in every 40 have severe asthma that needs the maximum available treatments advised in national asthma guidelines (known as the 'British Thoracic Society / Scottish Intercollegiate Guidelines Network British Guideline on the Management of Asthma'). Despite this, asthma is still inadequately controlled in about half of these patients and they are classed as having 'difficult asthma'. There maybe potential for improvement of the care and health of these patients through better use of medicines and greater input from pharmacists, but more research is needed.

The aim of the study is to measure the effects over six months of coordinated information and advice about medicines from hospital and community pharmacists on asthma control in patients with difficult asthma. The patients in the study (52 in total) will be recruited from adult patients attending a specialist difficult asthma clinic in a hospital.

Patients will be randomly chosen to have either an appointment with the specialist pharmacist (intervention group), or usual medical care (control group). Usual care will involve seeing the Consultant or Specialist Registrar (doctor) in the clinic. Patients in the intervention group will receive i) assessment and education on asthma, and review of their inhaler technique, from a hospital Advanced Clinical Pharmacist and ii) will also be referred for a medicines use review from their usual community pharmacist (chemist), to take place 1-2 months after their hospital clinic appointment. The Advanced Clinical Pharmacist will be working closely with the Consultant.

Results will be measured using methods that have been developed by experts in asthma and tested in previous research. Asthma control will be measured using Juniper's Asthma Control Questionnaire. Other measurements will cover quality of life, use of medication, use of healthcare resources, and inhaler technique.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of asthma
* Fulfil the criteria for difficult asthma (defined as persistent symptoms and/or frequent exacerbations despite treatment at step 4 or step 5 of the British TYhoracic Society / SIGN asthma guidelines 2011)
* Adult patients age between 18 and 70 years
* Able to speak, read and write in English
* All patients must have received their regular medication from the same Community Pharmacy for at least 3 months prior to their baseline visit
* Their community pharmacy must be registered with Leeds Primary Care Trust(PCT) to undertake targeted Medicines Use Reviews (tMURs).

Exclusion Criteria:

* Failure to meet the inclusion criteria
* Patient is not responsible for administering their own medications
* Patient is unlikely to be available for the 6-month follow-up period
* Failure to provide written informed consent
* Patient has had an MUR within the 12 months preceding the study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Improvement in Asthma Control, using Juiper's Asthma Control Questionnaire (ACQ). | 6 months